CLINICAL TRIAL: NCT02870010
Title: Chemoembolization of Non-resectable Non-metastatic Hepatocellular Carcinoma Using Embolization Microspheres (DC Bead™) Loaded With Idarubicin (Zavedos®): Phase 1 Study
Brief Title: Chemoembolization of Non-resectable Non-metastatic Hepatocellular Carcinoma Using Embolization Microspheres
Acronym: IDASPHERE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Boulin AOI 2009
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Localized Non-Resectable Adult Hepatocellular Carcinoma
MeSH Terms: interventions — Blood Specimen Collection; Chemoembolization, Therapeutic

ARMS (1):
- non-metastatic hepatocellular carcinoma (Experimental): * Radiation : Chemoembolization will take place in the Interventional Radiology room: the syringe, prepared at the pharmacy, will contain microspheres loaded with a defined dose of idarubicin. Then five millilitres of Visipaque® will be added to visualize the injection
  * Biological : blood samples (5 ml) will be taken
  Interventions: Biological: blood samples (5 ml) will be taken; Radiation: Chemoembolization

INTERVENTIONS:
Biological: blood samples (5 ml) will be taken — blood samples (5 ml) will be taken
Radiation: Chemoembolization — Chemoembolization will take place in the Interventional Radiology room: the syringe, prepared at the pharmacy, will contain microspheres loaded with a defined dose of idarubicin. Then five millilitres of Visipaque® will be added to visualize the injection

SUMMARY:
Chemoembolization is a recognized treatment strategy for hepatocellular carcinoma (HCC)

* classical chemoembolization consists in injecting an emulsion of an anticancer agent in Lipiodol® via the hepatic artery
* doxorubicin, an anthracycline, is the most frequently used drug in lipiodol chemoembolization (LCE)
* however, less than half of HCC respond favourably to classical lipiodol chemoembolization (LCE) with doxorubicin/Lipiodol®

In this trial, we propose to introduce in clinical practice a strategy based on idarubicin to achieve a more effective antitumor effect for the following reasons, recently pointed out by our team:

* idarubicin is an anthracycline that penetrates tumour cells more quickly and is more cytotoxic than doxorubicin on hepatocellular carcinoma cell lines
* idarubicin is injected in a solution of embolization microspheres of a diameter of (300-500µm), which all the progressive and controlled release of the anticancer drug, whereas the doxorubicin/Lipiodol® emulsion is unstable

ELIGIBILITY:
Inclusion Criteria:

-

Hepatocellular carcinoma(HCC) proven by cytology or histology or diagnosis according to the 2005 criteria of the American Association for the Study of Liver Diseases, (AASLD), which requires the presence of histological or unequivocal cirhosis and according to the size of nodules:

* nodule < 1 cm: increase in the size according to US scan every 3-4 months
* nodule between 1 and 2 cm: 2 concordant imaging techniques: CT-scan, MRI, contrast-enhanced US (CEUS); diagnosis of Hepatocellular carcinoma (HCC) in the presence of typical images (hypervascularized arterial + wash-out phase) with 2 imaging methods; in other cases, biopsy.
* nodule > 2 cm: CT-scan or MRI or CEUS (only 1 technique); diagnosis of Hepatocellular carcinoma (HCC) in the presence of hypervascularization associated with either a wash-out image or alphafoetoprotein> 200 µg/L; in other cases, biopsy.

  * A maximum of 3 nodules (Single-lobe disease - no limit to the number of nodules, in bilobar disease - a maximum of 3 nodules) distributed throughout the liver and detected by liver MRI with the injection of Gadolinium chelate, dating back less than 1 month. In cases of a contra-indication for MRI (pacemaker, metallic intra-ocular foreign body, certains cardiac valves et certains intra-cranial clips), a CT-scan with and without iodine-based contrast).
  * cases of cirrhosis: Child-Pugh stage A or B 7 without ascites, or icterus
  * WHO perfomance status 0, 1
  * Platelets > 50 000/mm3, Polynuclear neutrophils > 1000/mm3
  * Creatininemia < 150 µmol/l
  * Absence of heart failure (isotopic or US LVEF > 50%)
  * Age >18 years
  * Written informed consent

Exclusion Criteria:

* Patients able to undergo surgical resection or liver transplantation or local treatment with radio-frequency ablation
* Extra-hepatic metastases (lungs, bones, peritoneum...)
* Digestive haemorrhage dating back less than one month
* Patients on anticoagulants
* Portal thrombosis occurring in more than one segmental branch or hepatofugal flow on the Doppler
* Pregnant women
* Uncontrolled infection
* Hypersensitivity to anthracyclines
* Hypersensitivity to iodine contrast agents
* Patients under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-02; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Tolerance: toxicities will be defined according to the scale: National Cancer Institute - Common Toxicity Criteria for Adverse Events (NCI CTC AE v3.0) to determine the limiting dose | total duration of participation for a patient: 2 months
  Patients will be hospitalized for 3 days starting from the date of the chemoembolization and will then be followed regularly for 2 months from the date of the chemoembolization (clinical, biological and radiological surveillance).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de DIJON, Dijon, France